CLINICAL TRIAL: NCT02603965
Title: A Pilot Phase I Open Label Study of Cu-64-TP3805 PET Imaging for Detection of Prostate Cancer in Men Undergoing Radical Prostatectomy
Brief Title: Copper Cu 64 TP3805 PET in Detecting Cancer in Patients With Prostate Cancer Undergoing Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 13F.412; 2013-048 (Other: Thomas Jefferson University); NCI-2015-01533 (Registry Identifier: NCI Clinical Trials Reporting Program); JT 2479 (Other: JeffTrial Number)
Record Dates: First submitted 2015-11-04; First posted 2015-11-13 (Estimated); Last update posted 2025-05-02 (Actual); Status verified 2025-05

CONDITIONS: Prostate Adenocarcinoma; Stage IIB Prostate Cancer; Stage III Prostate Cancer; Stage IV Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Magnetic Resonance Spectroscopy; X-Rays

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Diagnostic (Cu 64 TP3805 PET/CT) (Experimental): Patients receive copper Cu 64 TP3805 IV and undergo PET/CT at 30 minutes and 2 hours post-injection. Patients then undergo radical prostatectomy within 1 to 3 weeks after scans.
  Interventions: Radiation: Copper Cu 64 TP3805; Procedure: Positron Emission Tomography; Procedure: Computed Tomography; Procedure: Radical Prostatectomy; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Radiation: Copper Cu 64 TP3805 — Given IV
  Other Names: Cu-64-TP3805
Procedure: Positron Emission Tomography — Undergo Cu-64-TP3805 PET(Positron Emission Tomography)/CT
  Other Names: Medical Imaging; Positron Emission Tomography Scan; PET SCAN; proton magnetic resonance spectroscopic imaging
Procedure: Computed Tomography — Undergo Cu-64-TP3805 PET/CT (Computed Tomography)
  Other Names: Computerized Axial Tomography; CT SCAN
Procedure: Radical Prostatectomy — Undergo radical prostatectomy
  Other Names: Prostatovesiculectomy
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This pilot phase I trial studies copper Cu 64 TP3805 (Cu-64-TP3805) positron emission tomography (PET)/computed tomography (CT) in detecting cancer in patients with prostate cancer undergoing surgery to remove the entire prostate and some of the tissue around it (radical prostatectomy). Many patients with benign lesions must undergo biopsy to test the lesion. Cu-64-TP3805 is a radioactive substance that attaches to cancer cells but not normal cells. PET/CT uses a scanner to make detailed, computerized pictures of areas inside the body where the radioactive substance is lighting up. Using Cu-64-TP3805 PET/CT scans and comparing them with cancer tissue obtained from surgery may help doctors learn whether Cu-64-TP3805 PET/CT can accurately detect prostate lesions and determine whether they are cancerous or benign, which may minimize the need for prostate biopsies.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the ability of Cu-64-TP3805 to detect prostate cancer (PC) within the prostate gland, as compared with whole mount step-sectioned surgical pathology of the prostate after radical prostatectomy.

OUTLINE:

Patients receive copper Cu 64 TP3805 intravenously (IV) and undergo PET/computed tomography (CT) at 30 minutes and 2 hours post-injection. Patients then undergo radical prostatectomy within 1 to 3 weeks after scans.

After completion of study, patients are followed up at 24 hours.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to provide signed informed consent and willingness to comply with protocol requirements
2. Biopsy confirmed presence of adenocarcinoma of the prostate gland
3. Have intermediate or high-risk PC as defined by >= T2b disease, or Gleason score >= 7 or prostate-specific antigen (PSA) >= 10 ng/dL
4. Scheduled to undergo radical prostatectomy with pelvic lymph node dissection (either open or robotic)
5. Agree to use an acceptable form of birth control for a period of 7 days after the Cu-64-TP3805 injection

Exclusion Criteria:

1. Participating would significantly delay the scheduled standard of care therapy
2. Administered a radioisotope within 10 physical half-lives prior to study drug injection
3. Have any medical condition or other circumstances that, in the opinion of the investigator, would significantly decrease obtaining reliable data, achieving study objectives or completing the study

Min Age: 21 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2013-08; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Detection rate of Cu-64 PET imaging of PC | Baseline (at time of surgery)
  The proportion of lesions detected with Cu-64 PET will be determined and compared with tumor maps derived from the whole mount step sectioned surgical pathology analysis of the radical prostatectomy specimen after surgery. 95% confidence intervals will be calculated. As a secondary analysis, a generalized estimating equations will be utilized to account for multiple lesions in an individual patient.
Incidence of adverse events | Up to 30 days post Cu-64-TP3805 injection procedure

CONTACTS AND LOCATIONS:
Overall Officials: Madhukar Thakur, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: Sidney Kimmel Cancer Center at Thomas Jefferson University, an NCI-Designated Cancer Center — http://www.KimmelCancerCenter.org
- See also: Thomas Jefferson University Hospital — http://hospitals.jefferson.edu/